CLINICAL TRIAL: NCT03584087
Title: Efficacy of Terlipressin Therapy in Acute Variceal Haemorrhage After Endoscopic Variceal Ligation: A Randomised Controlled Clinical Trial
Brief Title: Efficacy of Terlipressin Therapy in Acute Variceal Haemorrhage After EVL
Acronym: TEVL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Deba Prasad Dhibar, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEC/2018/000684
Record Dates: First submitted 2018-05-26; First posted 2018-07-12 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Acute Variceal Haemorrhage
Keywords: Terlipressin, Variceal Haemorrhage, EVL
MeSH Terms: interventions — Saline Solution; Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TG 0 (0Hr) (Placebo Comparator): TG0 will receive 10 ml of 0.9% normal saline (NS) IV bolus q 4 hourly in place of Terlipressin therapy after EVL.
  Interventions: Drug: Normal Saline
- TG 2 (48Hr) (Active Comparator): TG2 will receive Terlipressin (1mg, i.v. Bolus q 4 hourly) therapy for 48 hours after EVL .
  Interventions: Drug: Terlipressin
- TG 5 (120Hr) (Active Comparator): TG5 will receive Terlipressin (1mg, i.v. Bolus q 4 hourly) therapy for 120 hours after EVL .
  Interventions: Drug: Terlipressin

INTERVENTIONS:
Drug: Normal Saline — TG 0 (0Hr)
  Arms: TG 0 (0Hr)
Drug: Terlipressin — Duration of Terlipressin after EVL
  Arms: TG 2 (48Hr); TG 5 (120Hr)

SUMMARY:
Upper gastrointestinal (UGI) bleed of variceal origin is a common medical emergency. Prompt endoscopic variceal ligation (EVL) is therapeutic as well as diagnostic. Terlipressin, a vasopressin analog (intravenous, 2 mg q 4 hourly), is widely used promptly in any suspicious case of variceal haemorrhage (VH) before endoscopic procedure, along with volume and blood resuscitative measures. As per guideline, after EVL Terlipressin therapy (1 mg IV q 4 hourly) is continued for 2-5 day to prevent re-bleed. But the prolong use of Terlipressin is not completely safe as well as it is expensive also in resource constraint setting. At present there is no clinical trial available to prove the efficacy of post-EVL Terlipressin therapy in preventing re-bleed and mortality in cases of acute variceal haemorrhage. During the post marketing surveillance Terlipressin therapy has been found to be associated with life threatening complication like cardiac arrhythmia, myocardial ischemia, critical vasoconstriction of peripheral as well as internal organ leading to ischemia or gangrene, severe hyponatremia, hypertension, fluid overload and pulmonary oedema. So the justification of continuing Terlipressin therapy for 5 days after EVL is questionable, as haemostasis is primarily achieved by EVL and the risk versus benefit of Terlipressin therapy after EVL is still unknown. Continue IV Terlipressin therapy also prolongs in-hospital care causing further increase of health care burden. There is still lack of data of Terlipressin therapy, regarding its efficacy in preventing post-EVL re-bleed, mortality, adverse drug events and cost effectiveness. The investigator will study to evaluate the utility of Terlipressin therapy after EVL, in acute variceal haemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Irrespective of gender with age ≥ 18 years
* All the patients with endoscopy proven acute variceal haemorrhage (VH)
* Receiving Pre-EVL Terlipressin therapy
* EVL done within 24 hours of presentation
* Ready to give written informed consent

Exclusion Criteria:

* Patients with UGI bleed for more than 24 hours
* Not receiving pre-EVL Terlipressin therapy
* Pregnancy
* Past history of EVL
* Chronic kidney disease
* Patient's with EVL done beyond 24 hours of admission because of hemodynamic instability or encephalopathy
* Patients who are receiving blood thinners like anti-platelets, anti-coagulation agents within 4 weeks of presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with Early-Rebleed | 5 days
  To evaluate the efficacy of Terlipressin therapy to prevent re-bleed after EVL in acute variceal Haemorrhage (VH)
Number of participants with Rebleed | Within 2 Months
  To evaluate the efficacy of Terlipressin therapy to prevent re-bleed after EVL in acute variceal Haemorrhage (VH)
Early-Mortality | 7 days
  To evaluate the efficacy of Terlipressin therapy to prevent mortality after EVL in acute VH
Mortality | Within 2 Months
  To evaluate the efficacy of Terlipressin therapy to prevent mortality after EVL in acute VH

SECONDARY OUTCOMES:
Adverse drug events(ADE) | 5 days
  To evaluate ADE associated with Terlipressin therapy
Hospital Stay | Maximum 2 Months
  Duration of hospital Stay
Number of units of Blood transfusion during Hospital Stay | In hospital maximum upto 8 weeks
  Number of units of Blood transfusion during Hospital Stay
Cost of therapy | In hospital maximum upto 8 weeks
  Total cost of therapy during hospitalization
Complication | In hospital maximum upto 8 weeks
  Hepatic encephalopathy, need for mechanical ventilation, sepsis, shock, hospital acquired Pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Deba P Dhibar, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No